CLINICAL TRIAL: NCT06706674
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Study to Assess the Efficacy and Safety of Lumateperone in the Treatment of Irritability Associated With Autism Spectrum Disorder in Pediatric Patients 5 to 17 Years of Age
Brief Title: Multicenter Study of Lumateperone for the Treatment of Irritability Associated With Autism Spectrum Disorder (ASD) in Pediatric Patients
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-602
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Irritability Associated With Autism Spectrum Disorder
MeSH Terms: interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lumateperone high dose (Experimental): Lumateperone 42 mg for patients ages 13-17 years old
  Interventions: Drug: Lumateperone high dose
- Lumateperone low dose (Experimental): Lumateperone 21 mg for patients ages 13-17 years old
  Interventions: Drug: Lumateperone low dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lumateperone high dose — Lumateperone administered orally once daily
  Arms: Lumateperone high dose
Drug: Lumateperone low dose — Lumateperone administered orally once daily
  Arms: Lumateperone low dose
Drug: Placebo — Matching Placebo administered orally once daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study in pediatric patients aged 5 to 17 years with a primary diagnosis of irritability associated with Autism Spectrum Disorder (ASD) based on Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM-5-TR) and confirmed by the Kiddie Schedule for Affective Disorders and Schizophrenia Present and Lifetime Version (K-SADS-PL).

DETAILED DESCRIPTION:
The study will be conducted in 3 phases:

* Screening Period (up to 14 days) during which patient eligibility will be assessed.
* Double-blind Treatment Period (DBTP) (6 weeks) during which all patients will be randomized in a 1:1:1 ratio to receive either lumateperone high dose, lumateperone low dose, or placebo as a once daily dose.
* Safety Follow-up Period (1 week) during which all patients will return to the clinic for a safety follow-up (SFU) visit approximately 1 week after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have a legally authorized representative LAR (eg, parent or legal guardian) who is willing and able to be responsible for the safety and well-being of the patient, provide information about the patient's condition, and accompany the patient to study visits.
2. Able to provide consent as follows:

   1. The patient's LAR must provide written, informed consent.
   2. When developmentally appropriate based on Investigator judgment, the patient should provide written assent.
3. Male or female patients 5 to 17 years of age. Currently, only patients aged 13 to 17 years will be eligible for enrollment.
4. Meet Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition Text Revision (DSM-5-TR) primary diagnosis of ASD as confirmed by the Kiddie Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL);
5. ABC-I subscale score of >18 at Screening and Baseline;
6. CGI-S score > 4 with respect to irritability associated with ASD at Screening and Baseline.

Exclusion Criteria:

1. Has a primary psychiatric diagnosis other than ASD. Exceptions include:

   1. Attention Deficit Hyperactivity Disorder (ADHD). If a patient is taking medication(s) for ADHD, they must be on a stable treatment regimen of these medication(s) for 30 days prior to screening and the treatment regimen is expected to remain stable throughout the study. This must be confirmed by the Investigator and noted in the source records.
   2. Mild and moderate intellectual disability based on Investigator judgment and DSM-5 criteria (severe and profound intellectual disability are excluded).
2. History or current diagnosis of Rett syndrome or Fragile X syndrome;
3. In the opinion of the Investigator, the patient has a significant risk for suicidal behavior during their participation in the study or

   1. At Screening, the patient scores "yes" on Suicidal Ideation Items 3, 4, or 5 of the Columbia-Suicide Severity Rating Scale (CSSRS) within 6 months prior to Screening or, at Baseline, the patient scores "yes" on Suicidal Ideation Items 3, 4, or 5 since the Screening Visit;
   2. At Screening, the patient has had 1 or more suicidal attempts within the 2 years prior to Screening; or
   3. The patient is considered to be an imminent danger to themselves or others.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist - Irritability (ABC-I) | Week 6
  The ABC-I subscale contains 15 items which rate symptoms on a scale ranging from 0 (not at all a problem) to 3 (severe).

SECONDARY OUTCOMES:
Clinical Global Impression-Severity (CGI-S) | Week 6
  The CGI-S is a clinician-rated scale to assess a patient's overall mental health. The scale ranges from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Imperial, California
  - Clinical Site, Sacramento, California
  - Clinical Site, Sherman Oaks, California
  - Clinical Site, New Haven, Connecticut
  - Clinical Site, Hialeah, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Miami Gardens, Florida
  - Clinical Site, Miami Lakes, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Pompano Beach, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Lawrenceville, Georgia
  - Clinical Site, Naperville, Illinois
  - Clinical Site, Evansville, Indiana
  - Clinical Site, Indianapolis, Indiana
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Bloomfield Hills, Michigan
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Lincoln, Nebraska
  - Clinical Site, Orangeburg, New York
  - Clinical Site, Staten Island, New York
  - Clinical Site, The Bronx, New York
  - Clinical Site, Kinston, North Carolina
  - Clinical Site, Avon Lake, Ohio
  - Clinical Site, Oklahoma City, Oklahoma
  - Clinical Site, Charleston, South Carolina
  - Clinical Site, Austin, Texas
  - Clinical Site, Coppell, Texas
  - Clinical Site, Dallas, Texas
  - Clinical Site, Fort Worth, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, Richmond, Virginia
  - Clinical Site, Everett, Washington

IPD SHARING:
Plan to Share IPD: No